CLINICAL TRIAL: NCT05776537
Title: Assessment of Asthma Mimics Among Newly Diagnosed Bronchial Asthma Patients in Zagazig University Hospitals.
Brief Title: Assessment of Asthma Mimics Among Newly Diagnosed Bronchial Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZU-IRB # 6576/6-12-2020
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Asthma (Diagnosis)
Keywords: asthma, mimic diseases, spirometry
MeSH Terms: conditions — Asthma; Disease | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (1) confirmed bronchial asthma and group (2) bronchial asthma rule out (Other): After completing all the clinical, functional, radiologic, and endoscopic assessment, the patients were classified into two groups: Group (1) (89 patients) whose diagnosis confirmed to be bronchial asthma and group (2) (111 patients) with diagnoses other than bronchial asthma.
  Interventions: Device: Fibreoptic bronchoscopy

INTERVENTIONS:
Device: Fibreoptic bronchoscopy — different endoscopies used for confirmation of diagnosis
  Other Names: Upper Gastrointestinal (GI) endoscopy

SUMMARY:
The aim of the study was to identify the percentage of patients in whom the diagnosis of current asthma was confirmed or ruled out after clinical, spirometric assessment and utilizing all the possible investigations with a six month follow up period for both groups.

DETAILED DESCRIPTION:
The diagnosis of bronchial asthma relies on the existence of characteristic respiratory symptoms which are reversible and variable (diurnal and seasonal) with variable airflow limitation. Unfortunately, bronchial asthma may mimic different pulmonary and non-pulmonary diseases regarding their similar clinical presentations so accurate assessment is required to exclude other possible diagnosis before confirming the diagnosis of bronchial asthma.

There are various phenotypes of asthma as; atopic, non-atopic, and late-onset asthma, which may not be easily diagnosed in the community. Also, asthma may show intermittent versus a relapsing /remitting course, so it is difficult to be diagnosed by a single physician visit. Different studies have found that patients with bronchial asthma were treated empirically without full assessment either to ensure or exclude the asthma diagnosis.

Some symptoms as chest wheezes and breathlessness may be presented commonly in bronchial asthma and other mimic diseases as; chronic obstructive pulmonary disease, bronchiectasis, congestive heart failure, vocal cord disorders, hypersensitivity pneumonitis, endobronchial tumours, pulmonary embolism, aspiration syndromes, tracheal compression by a mediastinal mass and tracheomalacia. So, different physicians should put in mind those asthma mimics to be differentiated from asthmatic patients specially whose asthma symptoms are poorly controlled by anti- asthmatic medications.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients aged ≥ 18 years who had newly clinically diagnosed bronchial asthma (the diagnosis was achieved in the previous one year, to allow us to get the previous diagnostic reports) whether the diagnosis of asthma was initially made based on clinical assessment alone or both clinical and spirometric assessment. 2) Both sexes were included.

Exclusion Criteria:

* 1) Patients who were using long-term oral steroids that may mask the diagnosis; 2) unable to do spirometry or contra-indicated. 3) pregnancy. 4) Definite diagnosis of other chest diseases.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
the percentage of patients in whom the diagnosis of current asthma was confirmed or ruled out after clinical, spirometric assessment and utilizing all the possible investigations with a six month follow up period for both groups. | one month
  History of how patients were diagnosed as asthma: whether the diagnosis of asthma was initially made based on clinical assessment alone, or based on symptoms, physical findings, and diagnostic tests such as spirometry, reversibility test and peak expiratory flows.
  general and local chest examination. Spirometry The Asthma Control Questionnaire (ACQ-6) Sputum smear cytologic analysis Chest X-ray Electrocardiogram (ECG) and Echocardiography (ECHO). Chest computed tomography (Chest CT) Fibreoptic bronchoscopy with bronchial aspirate, lavage or biopsy if needed. Upper Gastrointestinal (GI) endoscopy and oesophageal motility assessment, Ear, Nose, and Throat (ENT) consultation and laryngoscopy Psychiatric consultation and psychotherapy, if indicated After completing all the previous clinical, functional, radiologic, and endoscopic assessment, A six month follow up period for both groups,

CONTACTS AND LOCATIONS:
Overall Officials: Samah M. Shehata, M.D., Principal Investigator — chest department, Zagazig university,Egypt
Locations (1):
- Chest Department,Faculty of Medicine, Zagazig, Egypt

REFERENCES:
- [Background] Blakey JD, Zaidi S, Shaw DE. Defining and managing risk in asthma. Clin Exp Allergy. 2014 Aug;44(8):1023-32. doi: 10.1111/cea.12334. PMID 24773229
- [Background] Aaron SD, Vandemheen KL, FitzGerald JM, Ainslie M, Gupta S, Lemiere C, Field SK, McIvor RA, Hernandez P, Mayers I, Mulpuru S, Alvarez GG, Pakhale S, Mallick R, Boulet LP; Canadian Respiratory Research Network. Reevaluation of Diagnosis in Adults With Physician-Diagnosed Asthma. JAMA. 2017 Jan 17;317(3):269-279. doi: 10.1001/jama.2016.19627. PMID 28114551